CLINICAL TRIAL: NCT05160467
Title: Bio Electrical Impedance Analysis to Monitor Fluid Status During Deresuscitation Strategy in Continuous Renal Replacement Therapy: a Proof of Concept Study
Brief Title: Bio Electrical Impedance Analysis to Monitor Fluid Status During Deresuscitation Strategy in Continuous Renal Replacement Therapy
Acronym: UF BIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 532
Record Dates: First submitted 2021-11-22; First posted 2021-12-16 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Fluid Overload
Keywords: bio electrical impedance analysis; fluid overload; deresuscitation strategy; net ultra filtration
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Deresuscitation cohort: Patients with fluid overload (defined by a cumulative fluid balance > 5%), stable hemodynamic (defined by Norepinephrine equivalent < 0.5µg/kg/min and nor clinical nor biological sign of hypoperfusion) and continuous renal replacement therapy. All these patients benefit in our service from a protocol directed, perfusion based deresuscitation strategy with a 2mL/kg/h net ultra filtration to induce negative fluid balance and correct fluid overload. If hypoperfusion occurs, the net ultra filtration is stopped; if pulmonary oedema or right ventricular dysfunction occurs, the net ultra filtration is set to 3mL/kg/h.
  We carried out at day 0, 1,3 and 5 bio electrical impedance analysis with an eight polar multifrequency bio impedance monitor (InBody S10), and monitor cumulative fluid balance with our prescription software and daily weight assessment.
  Interventions: Diagnostic Test: Segmental multi-frequency bio electrical impedance analysis

INTERVENTIONS:
Diagnostic Test: Segmental multi-frequency bio electrical impedance analysis — A segmental (eight-polar) multi-frequency bio electrical impedance analysis (Inbody S10, Seoul, Korea) is carried out at the initiation of the deresuscitation strategy, at day 1, 3 and 5, in lying posture with touch type electrodes. Raw and derived parameters are recorded. The measurement is performed 5 times for the first measurement and then one time at day 1, 3 and 5.
  Measurement error is defined by the manufacturer as: reversed Impedance in different segment all between 5-500kHz; impedance over 50Ω in trunk, or over 700Ω in limb; sudden drop of impedance in trunk (more than 10Ω), or in limb (more than 50Ω). If it occurs, measurement is carried out three times maximum after solving potential technical issues to obtain a valid analysis.

SUMMARY:
Fluid overload is a poor prognostic factor in patients undergoing continuous renal replacement therapy in critical care. A strategy of active fluid removal by net ultrafiltration (UFnet) is one of the means to correct it. However, fluid overload is difficult to quantify: weight variations or cumulative fluid balance are easy to use but imprecise and not concordant markers, while reference methods such as isotope dilution are not adapted to daily practice.

Bio electrical impedance analysis (BIA) is used to estimate body composition, including hydration. It is a non-invasive, rapid and painless measurement. It is commonly used in chronic intermittent haemodialysis to estimate dry weight and guide fluid removal, with a demonstrated impact on blood pressure control. This analysis is feasible in the ICU. Fluid overload as defined by BIA correlates with mortality, most notably in acute renal failure and during continuous renal replacement therapy.

We routinely perform multifrequency segmental BIA (InBody S10, Seoul, Korea) in patients with fluid overload in our intensive care department. Since February 2021, we have implemented a protocol to systematically correct fluid overload by inducing negative fluid balance with UFnet in a manner appropriate to tissue perfusion. In this context, we systematically perform a BIA analysis on the day of the beginning of the fluid balance negativation and then every 48 hours during the first five days.

We would like to evaluate the relevance of BIA monitoring in these patients by comparing it to other parameters of evaluation of the volume status usually used.

ELIGIBILITY:
Inclusion Criteria:

* Age higher than 18
* Protocol directed deresucitation strategy with net ultrafiltration during continuous renal replacement therapy
* Bioelectrical impedance analysis available for the day of the initiation of the deresuscitation strategy and at day 5" -> "At least two bioelectrical impedance analysis available during the first 5 days of the initiation of the deresuscitation strategy".

Exclusion Criteria:

* Left ventricular assist device
* Patient opposition to the use of his health data
* Invalid bioelectrical impedance analysis
* Advanced directives to withhold or withdraw life-sustaining treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fluid overload (defined by a cumulative fluid balance > 5%), stable hemodynamic (defined by Norepinephrine equivalent < 0.5µg/kg/min and nor clinical nor biological sign of hypoperfusion) and continuous renal replacement therapy. All these patients benefit in our service from a protocol directed, perfusion based deresuscitation strategy with net ultra filtration to induce negative fluid balance.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between changes in extracellular water volume estimated by BIA and cumulative fluid balance between day 0 and day 5 (mL). | Coefficient correlation between the variation from day 0 to day 5 of extra cellular water and cumulative fluid balance
  The extra cellular water is a volumetric value, given automatically by the InBody S10 device. The cumulative fluid balance at day 5 is the sum of the daily fluid balances between day 0 and day 5.
  Definition of the fluid balance = inputs - outputs :
  * Inputs = total cumulative volume of: parenteral medication; enteral and parenteral nutrition; maintenance fluid; blood products; fluid bolus therapy
  * Outputs = total cumulative volume of: diuresis; losses to drain; net ultra filtration

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital cardiologique Louis Pradel Groupe Hospitalier Est, Bron, France